CLINICAL TRIAL: NCT03140436
Title: Clinical Comparison of the Stain Removal Efficacy of Two Air Polishing Powders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015/DT035
Record Dates: First submitted 2017-04-26; First posted 2017-05-04 (Actual); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Stain Removal Efficacy
Keywords: stain removal efficacy, air polishing powder

STUDY DESIGN:
Intervention Model Description: This study was designed as a double-blind, randomized split-mouth design.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Each group received treatment through a different operator (one operator per one group). Each patient was randomized using sealed envelopes according to treatment side (right or left) using powder grain size 65 µm or 40 µm. The patients and operators were blinded from the type of the powder.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sodium bicarbonate powders (65 µm) (Experimental): sodium bicarbonate powders with grain size 65 µm
  Interventions: Drug: sodium bicarbonate powders with grain size 65 µm
- sodium bicarbonate powders (40 µm) (Experimental): sodium bicarbonate powders with grain size 40 µm
  Interventions: Drug: sodium bicarbonate powders with grain size 40 µm

INTERVENTIONS:
Drug: sodium bicarbonate powders with grain size 65 µm — sodium bicarbonate powders with grain size 65 µm
  Other Names: sodium bicarbonate powders
  Arms: sodium bicarbonate powders (65 µm)
Drug: sodium bicarbonate powders with grain size 40 µm — sodium bicarbonate powders with grain size 40 µm
  Other Names: sodium bicarbonate powders
  Arms: sodium bicarbonate powders (40 µm)

SUMMARY:
This study was designed to find out the stain removal efficacy and also, to find out the operators and patients opinion when use or receive treatment with both air polishing powders.

DETAILED DESCRIPTION:
Using air polishing with sodium bicarbonate powders with grain size 65 µm provides efficacy in the removal of dental stains but it can cause gingival trauma if used towards the gingiva. Since having big size particles is uncomfortable, the current recommendation according to literature is to use a smaller grain size (40 µm) that results in more patient comfort. However, the efficacy of small grain size on stain removal has not been studied adequately. This study aimed to compare the stain removal efficacy between sodium bicarbonate powders with grain size 65 µm and 40 µm and also to evaluate patient's acceptance after treatment and operator's opinion after using both air polishing powders.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects who aged over 18 years old.
2. Subjects who have healthy periodontal health or gingivitis.
3. At least 3 upper teeth (anterior, premolar and molar) are presented on both side (right & left side), which will be refer as index teeth, that did not present with any gingival recession, cervical abrasion and/or abfraction, caries, restoration or orthodontic appliance.
4. Intrinsic stain is not present.
5. Index teeth are presented with extrinsic stain with individual Lobene score scored 2 or above.

Exclusion Criteria:

1. Pregnancy or current breastfeeding mother.
2. Allergy to sodium bicarbonate or the aroma of the powder

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
The time required for complete removal of extrinsic stains | 2 hr
  Comparison of the time required for the complete removal of extrinsic stains by sodium bicarbonate powders with a grain size of 65 µm and 40 µm

SECONDARY OUTCOMES:
Patient acceptance | 2 hr
  The answers from the questionnaires about the clinical impressions of patients after treatment with sodium bicarbonate powders with a grain size of 65 µm and 40 µm
Operator opinion | 2 hr
  The answers from the questionnaires about the operators' opinions after using of sodium bicarbonate powders with a grain size of 65 µm and 40 µm

CONTACTS AND LOCATIONS:
Overall Officials: Kanyawat Rattanasuwan, Study Director — Mahidol University
Locations (1):
- Kanyawat Rattanasuwan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No